CLINICAL TRIAL: NCT04757350
Title: Objective Visual Quality Analysis System is Used to Evaluate the Effect of Cataract Surgery and Manage Postoperative Complications
Brief Title: Objective Visual Quality Analysis System is Used in Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yukan Huang, professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: YKHYK2020
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cataract: Research subjects should meet the following criteria: Signed and dated informed consent form Commitment to abide by the research procedures and cooperate with the implementation of the whole process of research 18-90-year-old cataract patients or patients after cataract surgery
  Interventions: Other: Observational research, not applicable

INTERVENTIONS:
Other: Observational research, not applicable — Observational research, not applicable

SUMMARY:
The Objective Visual Quality Analysis System (OQAS) is a new inspection technology used to objectively assess the visual quality of the human eye. The investigators use this advanced technology to evaluate and follow up cataract patients before and after surgery, and observe the incidence, severity, and treatment effects of postoperative complications such as postoperative complications, and analyze the severity and artificial The influence of lens type, postoperative time, systemic diseases and other factors on the effect of cataract surgery, in order to discover the key factors that affect the effect of cataract surgery and the management of complications, and provide a useful reference for improving the level of cataract prevention and treatment in China

DETAILED DESCRIPTION:
The Objective Visual Quality Analysis System (OQAS) is a new inspection technology used to objectively assess the visual quality of the human eye. It can detect the impact of ocular refractive system diseases on the objective visual quality of patients. It is currently mainly used to assess the progress of cataracts and help selection the timing of surgery has achieved good clinical results. Before the emergence of OQAS, the rating of cataracts largely relied on the subjective experience of physicians, and OQAS could accurately assess the effects of cataracts on the visual quality of the human eye by quantitatively detecting the light scattering index (OSI) of the refractive medium of the human eye. The impact provides a quantitative evaluation basis for the diagnosis and treatment of cataract and research. However, the application of OQAS in cataract surgery effect evaluation and postoperative complications management is still lacking. After cataract surgery, although the cloudy lens nucleus and cortex have been removed, the original refractive error, vitreous opacity, postoperative posterior capsule folds, posterior dysfunction and many other factors may still affect the objective of the human eye visual quality, and ordinary visual inspection is difficult to find this effect . In addition, preoperative OSI and other indicators of cataract, as an exposure factor, may affect the incidence of postoperative complications, such as after-cataract, macular edema, etc. It is worthy of further study. The application of OQAS can accurately assess the improvement of objective visual quality after cataract surgery, and find and remove other factors that affect OSI. In addition, for one of the most common complications after cataract surgery-after-onset disorder, there is no uniform rating standard in the academic circles, and OQAS can provide objective data for the rating of after-onset disorder, so as to provide information on the postoperative complications such as late-onset disorder. Provide reference for the management of . The research team intends to use OQAS to evaluate and follow up cataract patients before and after surgery, and observe the incidence, severity, and treatment effects of postoperative complications such as after-cataract, analyze the severity of cataract or after-cataract, and intraocular lens The influence of factors such as type, postoperative time, systemic disease on the effect of cataract surgery. We will also rate the posterior disorder based on OSI, and examine the effects and risks of different grades of posterior disorder after laser capsulotomy and other treatments, in order to use OQAS to better guide cataract surgery and postoperative complications management.

ELIGIBILITY:
Inclusion Criteria:

1. Cataract patients aged 18-90 or patients after cataract surgery；
2. Signed and dated informed consent；
3. Commit to abide by the research procedures and cooperate with the implementation of the whole process research

Exclusion Criteria:

1. Obvious conjunctivitis；
2. Obvious corneal epithelial punctate staining, corneal epithelial shedding；
3. Keratitis；
4. Uveitis；
5. Corneal scar；
6. Severe vitreous opacity or hemorrhage；
7. Other situations deemed unsuitable for inclusion in this study after evaluation by ophthalmologists.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Union Hospital Eye Clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from visual acuity at 6 months | 6 months
  VA after cataract surgery 1 week、1month、3month、6month
Change from Objective Scatter Index at 6 months | 6 months
  OSI after cataract surgery 1 week、1month、3month、6month
Change from Contrast Sensitivity at 6 months | 6 months
  CS after cataract surgery 1 week、1month、3month、6month
Change from Patient Satisfaction Scale at 6 months | 6 months
  Patient Satisfaction Scale after cataract surgery 1 week、1month、3month、6month.The minimum values is 0 and maximum values is 100.100 points mean the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: yukan huang, professor, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Wuhan, Hubei, China